CLINICAL TRIAL: NCT02360449
Title: Social Motivation Intervention for Children With Autism Spectrum Disorder: Improving Peer Initiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grace Gengoux, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31420
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Pivotal Response Treatment; Applied Behavior Analysis; Peer Initiation; Social Skills Group
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait List (No Intervention)
- Social Initiation Motivation Intervention (Experimental)
  Interventions: Behavioral: Social Initiation Motivation Intervention

INTERVENTIONS:
Behavioral: Social Initiation Motivation Intervention — The SIMI approach under investigation uses behavioral strategies based in Applied Behavior Analysis and Pivotal Response Treatment to motivate children with ASD to initiate to peers. The adult arranges the play environment in order to promote cooperation and facilitates frequent prompting and reinforcement from peers, thereby enhancing the reward value of peer interactions.
  Other Names: Pivotal Response Treatment
  Arms: Social Initiation Motivation Intervention

SUMMARY:
The purpose of this study is to investigate whether a social initiation motivation intervention (SIMI) focused on training children with ASD to initiate to peers during structured play activities will result in more frequent initiations to typically developing peers during free play. The SIMI approach under investigation uses behavioral strategies based in Applied Behavior Analysis and Pivotal Response Treatment to motivate children with ASD to initiate to peers. Children with ASD will be randomly assigned to either the SIMI or a waiting list. Treatment will be provided for 8 weeks in the context of a weekly social skills group.

ELIGIBILITY:
Inclusion Criteria:

1. age 4.0 to 6.11 years;
2. diagnosis of Autism Spectrum Disorder
3. without intellectual disability
4. stable community treatments four weeks before and throughout the trial.

Exclusion criteria:

1. diagnosed severe psychiatric or genetic disorder or medical problem;
2. severe disruptive behavior that would interfere with peer interactions

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Initiation Frequency (observational rating of the frequency of child initiations to peers measured from video recording during free play sessions) | 8 weeks
  The primary measure is an observational rating of the frequency of child initiations to peers measured from video recording during free play sessions at baseline and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Gengoux, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Result] Gengoux GW, Schwartzman JM, Millan ME, Schuck RK, Ruiz AA, Weng Y, Long J, Hardan AY. Enhancing Social Initiations Using Naturalistic Behavioral Intervention: Outcomes from a Randomized Controlled Trial for Children with Autism. J Autism Dev Disord. 2021 Oct;51(10):3547-3563. doi: 10.1007/s10803-020-04787-8. Epub 2021 Jan 2. PMID 33387236
- See also: Published primary trial results (Stanford Medical Library link) — https://lane.stanford.edu/view/pubmed/33387236